CLINICAL TRIAL: NCT04483258
Title: Cross-over Analysis of Sevoflurane Insufflation and Intravenous Sedation for Radiotherapy in Pediatric Patients
Brief Title: Sevoflurane Insufflation vs Intravenous Sedation for Radiotherapy in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: E1-20-884
Record Dates: First submitted 2020-07-18; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Pediatric Sedation; Radiotherapy; Inhalation Anesthesia
Keywords: insufflation sedation; intravenous sedation; radiotherapy anesthesia; pediatric sedation

STUDY DESIGN:
Intervention Model Description: Sevoflurane insufflation and intravenous sedation will be applied to the patients by changing them sequentially during each radiotherapy session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation with Insufflation (Active Comparator): Sedation induction via oxygen mask %8 sevoflurane and reducing %3 concentration after rediotherapy start
  Interventions: Procedure: Sedation with sevoflurane insufflation
- İntravenous sedation (Active Comparator): Midazolam+ Ketamine sedation
  Interventions: Procedure: intravenous sedation

INTERVENTIONS:
Procedure: Sedation with sevoflurane insufflation — Induction with %8sevoflurane after adequate sedation reducing %3
  Arms: Sedation with Insufflation
Procedure: intravenous sedation — midazolam +ketamine + atropine
  Arms: İntravenous sedation

SUMMARY:
aim of this cross-over study is to compare sedation with insufflated sevoflurane and intravenous sedation for pediatric radiotherapy patients

DETAILED DESCRIPTION:
aim of this cross-over study is to compare sedation with insufflated sevoflurane and intravenous sedation for pediatric radiotherapy(RT) patients in terms of success of the procedure (continuous completion of the RT session by providing inactivity) and complications such as desaturation, hypoventilation, airway spasm, bradycardia, tachycardia In addition, we aimed to investigate the incidence of anesthesia complications in RT patients and possible related factors with complications.

ELIGIBILITY:
Inclusion Criteria:

* undergoing radiotherapy session

Exclusion Criteria:

* family refusal
* chronic nausea and vomiting
* apnea history, pneumonia, asthma, bronchiolitis etc. respiratory tract infection or diseases
* cardiac disease
* kidney failure
* liver failure
* anticipated difficult airway
* metabolic diseases
* neurological or muscular diseases.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
number of the successful radiotherapy sessions | during radiotherapy session
  succesful: radiotherapy session without interruption unsuccesful: radiotherapy session with any interruption
number of interruptions | during radiotherapy session
  number of interruptions related to inadequate sedation and patient's movement in radiotherapy session
PSSS | during radiotherapy session
  5:Patient is moving 4: gentle immobilization for positioning. 3: do not require restraint to stop movement during the procedure. 2: Quiet (asleep or awake), not moving during procedure
  1: Deeply asleep with normal vital signs, but requiring airway intervention 0: Sedation associated with abnormal physiologic parameters that require acute intervention

SECONDARY OUTCOMES:
sPO2 | during radiotherapy session
  peripheral oxygen saturation
HR | during radiotherapy session
  Heart Rate

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytac, Principal Investigator — Ankara City Hospital Anesthesiology Department
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No